CLINICAL TRIAL: NCT03375385
Title: Effect of Dexmedetomidine Versus Propofol on the Onset and Recovery of Sedation in Stereotactic Brain Biopsy A Comparative Study
Brief Title: Dexmedetomidine Versus Propofol for Sedation in Stereotactic Brain Biopsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ghada M.Samir, assistant professor of anaesthesia and intensive care, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU R44/ 2017
Record Dates: First submitted 2017-12-04; First posted 2017-12-18 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Adverse Effects in the Therapeutic Use of Other and Unspecified Agents Primarily Acting on the Respiratory System
MeSH Terms: interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hemodynamic parameters (Other)
  Interventions: Drug: dexmedetomidine/ propofol
- Ramsay sedation score (Other)
  Interventions: Drug: dexmedetomidine/ propofol
- Intraoperative side effects (Other)
  Interventions: Drug: dexmedetomidine/ propofol
- recovery of sedation (Other)
  Interventions: Drug: dexmedetomidine/ propofol

INTERVENTIONS:
Drug: dexmedetomidine/ propofol — The loading and infusion doses of dexmedetomidine hydrochloride and 1% propofol were calculated according to the patient's body weight and diluted to a 10 ml volume (labeled as loading-1 and loading-2) and a 50 ml volume (labeled as infusion-1 and infusion-2).

SUMMARY:
Pre-operative anxiety leads to higher sympathetic stimulation. Propofol in the main drug used during interventional or imaging techniques that need sedation. Also, dexmedetomidine causes sedation, analgesia, sympatholytic properties, without respiratory depression.In stereotactic brain biopsy; patient discomfort due to drilling a hole through the skull and the advancement of the biopsy needle make the patient in need for good sedation and analgesia.

ELIGIBILITY:
Inclusion criteria:

Patients with:

* brain secondaries from the lung/breast/pancreas
* tuberculoma
* pyogenic abscess
* intra-axial supratentorial space occupying lesion with or without hydrocephalus *an average duration of the procedure 1- 2hr 30 min
* an available caregiver for overnight observation
* patient relative proximity to the hospital Exclusion criteria

Patients with:

* morbid obesity (body mass index >35 kg/m2)
* significant comorbidities (a known history of hepatic disease, renal dysfunction, hypertension, and chronic pain)
* history of drug or alcohol abuse
* an allergic reaction to one of the study medications
* anticipated difficult airway
* uncontrolled epilepsy
* poor neurological status
* neuropsychological unsuitability taking psychotropic drugs (benzodiazepines and barbiturates)
* patients with brain stem lesions (vital areas of brain)
* un-cooperative
* refusing adults
* patients with ventricular drain
* already inpatient
* Intubated patients and those who had a prior craniotomy .

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
the sedation characteristics | 4 hours
  Ramsay sedation score

IPD SHARING:
Plan to Share IPD: No